CLINICAL TRIAL: NCT03338036
Title: The Effectiveness of Neurofeedback and Heart Rate Variability Biofeedback for Individuals With Long-term Post-concussive Symptoms
Brief Title: The Effectiveness of Biofeedback for Individuals With Long-term Post-concussive Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: Parkwood Hospital, London, Ontario (Other)
Responsible Party: Principal Investigator, James Dickey, Sponsor-Investigator, Western University, Canada
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Western University REB 109760
Record Dates: First submitted 2017-11-03; First posted 2017-11-09 (Actual); Results first posted 2020-06-04 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-07

CONDITIONS: Post-Concussion Syndrome
Keywords: Concussion; Post-Concussion Syndrome; Biofeedback; Heart Rate Variability; Neurofeedback
MeSH Terms: conditions — Post-Concussion Syndrome; Brain Concussion | interventions — Neurofeedback

STUDY DESIGN:
Intervention Model Description: This study will include two intervention arms and two control arms. The intervention arms will include 1) heart rate variability biofeedback, 2) a combination of heart rate variability biofeedback and neurofeedback. The control arms will be 1) age-matched post-concussive individuals and 2) age-matched individuals who have not been diagnosed with a concussion in the last two years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Heart Rate Variability/Neurofeedback (Experimental): Participants in this arm of the study will receive HRV biofeedback and neurofeedback. HRV biofeedback will occur twice daily, using an android device and application. Additionally, three times per week they will have one-hour long neurofeedback sessions.
  Interventions: Device: Heart Rate Variability Biofeedback; Device: Neurofeedback
- Post-Concussed Control Group (No Intervention): Age-matched, previously concussed individuals that have completed the same concussion rehabilitation program (Brain Ex 90) will be recruited for this arm.
- Non-Concussed Control Group (No Intervention): Age-matched individuals who have not been diagnosed with a concussion in the previous two years

INTERVENTIONS:
Device: Heart Rate Variability Biofeedback — HRV biofeedback constitutes initial training with the android device and application, and HRV training performed at home. This training will occur twice daily, and each session will take five minutes.
  Arms: Heart Rate Variability/Neurofeedback
Device: Neurofeedback — LORETA Z-Score neurofeedback training will occur three times per week with a trained study investigator.
  Arms: Heart Rate Variability/Neurofeedback

SUMMARY:
Most concussions resolve within 7-10 days, but approximately 40% of individuals do not fully recover and suffer from persistent post-concussive symptoms. This 8-week intervention study will evaluate the efficacy of heart rate variability (HRV) biofeedback and neurofeedback on reducing the number and severity of concussion symptoms.

DETAILED DESCRIPTION:
40% of minor head injuries are diagnosed with post-concussion syndrome 3 months after injury (Ingebrigtsen, Waterloo, Marup-Jensen, Attner, & Romner, 1998). These individuals have persistent symptoms after completing conventional rehabilitation programs. Persistent post-concussion symptoms not only decrease quality of life (Ingebrigtsen et al, 1998), but also impair cognitive and motor performance and increase the likelihood of impaired driving performance (Preece, Horswill, & Geffen, 2010) and motor vehicle accidents (Bivona et al, 2012). While case reports indicate that biofeedback can reduce the number and severity of post-concussive symptoms (Lagos, Thompson, & Vaschillo, 2013; Thompson, Thompson, Reid-Chung, & Thompson, 2013), no studies have systematically evaluated these biofeedback treatment programs.

HRV biofeedback works by displaying beat-to-beat heart rate data to the participant, and through operant conditioning with breathing techniques, the participant learns to control their HRV (Lehrer & Gevirtz, 2014). This results in an increase in parasympathetic (PNS) activity and decrease in sympathetic (SNS) activity, which leads to reduced anxiety, and increased focus and concentration (Lagos, Bottiglieri, Vaschillo, & Vaschillo, 2012). Neurofeedback works in a similar fashion, except it monitors brain wave power, frequency, and connectivity using quantitative electroencephalogram (EEG). Brain functioning is displayed while playing an electronic game, and the participant learns through operant conditioning to increase the amplitude of desired EEG frequencies, such as low beta waves that are associated with active problem solving, usually while simultaneously decreasing the amplitudes of undesired EEG frequencies (Conder & Conder, 2014).

This will be an eight-week intervention where participants suffering from long-term post-concussion symptoms will be recruited using email from the cohort of individuals that have been discharged after completing a concussion rehabilitation protocol (BrainEx90) at Parkwood Institute in London, Ontario. Non-concussed control participants will be recruited using posters. Participants will complete pre, mid, and post-intervention driving simulation tasks, electrocardiogram and HRV measures, and subjective questionnaires. These will be utilized to evaluate the effectiveness of HRV biofeedback and neurofeedback in this difficult to treat population.

ELIGIBILITY:
Inclusion Criteria:

Participants in HRV and the HRV/Neurofeedback intervention arms, and the post-concussion control arm:

1. Previously suffered a clinically diagnosed concussion
2. Participated in, completed, and have been discharged from the BrainEx90 outpatient concussion rehabilitation program at Parkwood Institute
3. Continued post-concussive symptoms
4. 18 years of age or older
5. Access to transportation
6. Capable of utilizing hand-held technology (ie. cell phone, tablet, etc.)
7. Holds a valid Driver's License
8. English speaking

Participants in the non-concussed control arm:

1. 18 years of age or older
2. Holds a valid driver's license
3. English speaking
4. Has not suffered a concussion in the last two years

Exclusion Criteria:

All participants:

1. Any heart disease, pacemaker, abnormal heartbeat patterns, coronary artery disease, or bypass surgery
2. Any mental health disorder that would interfere with participation in the study
3. Under 18 years of age
4. Unable to provide written informed consent or complete questionnaires due to language or cognitive difficulties
5. Inability to operate a motor vehicle
6. Inability to look at a digital screen for 30 minutes

Participants in the non-concussed control arm:

1. Suffered a concussion in the last two years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James P Dickey, PhD, Principal Investigator — Western University
Locations (1):
- University of Western Ontario, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Each participant will be identified with a code (eg. PCS001) that correlates to his or her addition to the study. The master sheet will be the only document that contains the decoding system, and will be stored in a locked filing cabinet. All other data will be labeled using the participant's identification code.
  Neurophysiological data sent to Evoke Neuroscience will not contain any personal identifiers. Data sent between Evoke Neuroscience and Western University is sent in a secure file transfer. All other de-identified data stored on a Western University hard drive is within a secure university network (J drive).

REFERENCES:
- [Background] Bivona U, D'Ippolito M, Giustini M, Vignally P, Longo E, Taggi F, Formisano R. Return to driving after severe traumatic brain injury: increased risk of traffic accidents and personal responsibility. J Head Trauma Rehabil. 2012 May-Jun;27(3):210-5. doi: 10.1097/HTR.0b013e31822178a9. PMID 21829135
- [Background] Conder RL, Conder AA. Heart rate variability interventions for concussion and rehabilitation. Front Psychol. 2014 Aug 13;5:890. doi: 10.3389/fpsyg.2014.00890. eCollection 2014. PMID 25165461
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Fisk GD, Schneider JJ, Novack TA. Driving following traumatic brain injury: prevalence, exposure, advice and evaluations. Brain Inj. 1998 Aug;12(8):683-95. doi: 10.1080/026990598122241. PMID 9724839
- [Background] Gevensleben H, Holl B, Albrecht B, Schlamp D, Kratz O, Studer P, Rothenberger A, Moll GH, Heinrich H. Neurofeedback training in children with ADHD: 6-month follow-up of a randomised controlled trial. Eur Child Adolesc Psychiatry. 2010 Sep;19(9):715-24. doi: 10.1007/s00787-010-0109-5. Epub 2010 May 25. PMID 20499120
- [Background] Ingebrigtsen T, Waterloo K, Marup-Jensen S, Attner E, Romner B. Quantification of post-concussion symptoms 3 months after minor head injury in 100 consecutive patients. J Neurol. 1998 Sep;245(9):609-12. doi: 10.1007/s004150050254. PMID 9758300
- [Background] Lagos, L., Bottiglieri, T., Vaschillo, B., & Vaschillo, E. (2012). Heart Rate Variability Biofeedback for Postconcussion Syndrome: Implications for Treatment. Biofeedback, 40(4), 150-153. doi:10.5298/1081-5937-40.4.05
- [Background] Lagos, L., Thompson, J., & Vaschillo, E. (2013). A Preliminary Study: Heart Rate Variability Biofeedback for Treatment of Postconcussion Syndrome. Biofeedback, 41(3), 136-143. doi:10.5298/1081-5937-41.3.02
- [Background] Lehrer PM, Gevirtz R. Heart rate variability biofeedback: how and why does it work? Front Psychol. 2014 Jul 21;5:756. doi: 10.3389/fpsyg.2014.00756. eCollection 2014. PMID 25101026
- [Background] Milleville-Pennel I, Pothier J, Hoc JM, Mathe JF. Consequences of cognitive impairments following traumatic brain injury: Pilot study on visual exploration while driving. Brain Inj. 2010;24(4):678-91. doi: 10.3109/02699051003692159. PMID 20235770
- [Background] Munivenkatappa A, Rajeswaran J, Indira Devi B, Bennet N, Upadhyay N. EEG Neurofeedback therapy: Can it attenuate brain changes in TBI? NeuroRehabilitation. 2014;35(3):481-4. doi: 10.3233/NRE-141140. PMID 25238859
- [Background] Preece MH, Horswill MS, Geffen GM. Driving after concussion: the acute effect of mild traumatic brain injury on drivers' hazard perception. Neuropsychology. 2010 Jul;24(4):493-503. doi: 10.1037/a0018903. PMID 20604623
- [Background] Thompson, M., Thompson, L., Reid-Chung, A., & Thompson, J. (2013). Managing Traumatic Brain Injury: Appropriate Assessment and a Rationale for Using Neurofeedback and Biofeedback to Enhance Recovery in Postconcussion Syndrome. Biofeedback, 41(4), 158-173. doi:10.5298/1081-5937-41.4.07

RESULTS

PARTICIPANT FLOW:
Groups:
- Heart Rate Variability Biofeedback: Participants in this arm of the study will only receive HRV biofeedback. This constitutes initial training with the android device and application, and HRV training performed at home. This training will occur twice daily, and each session will take five minutes. Participants in this arm will meet with the co-investigator bi-weekly to review progress and express feedback.
  Heart Rate Variability Biofeedback: HRV biofeedback constitutes initial training with the android device and application, and HRV training performed at home. This training will occur twice daily, and each session will take five minutes.
Period: Overall Study
Arm/Group | Heart Rate Variability Biofeedback | Heart Rate Variability/Neurofeedback | Post-Concussed Control Group | Non-Concussed Control Group
Started | 0 | 11 | 12 | 8
Completed | 0 | 7 | 9 | 8
Not Completed | 0 | 4 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Given our low recruitment rate, we abandoned one arm of the study; the Heart Rate Variability Biofeedback arm was abandoned.
Groups:
- Total: Total of all reporting groups
Arm/Group | Heart Rate Variability Biofeedback | Heart Rate Variability/Neurofeedback | Post-Concussed Control Group | Non-Concussed Control Group | Total
Number analyzed (Participants) | 0 | 7 | 9 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 48.6 (13) | 54.6 (7.6) | 50.1 (15.5) | 51.21 (12.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 4 | 6 | 4 | 14
  Male |  | 3 | 3 | 4 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada |  | 7 | 9 | 8 | 24
RPQ [Mean (Standard Deviation); unit: units on a scale] — The Rivermead Post-Concussion Questionnaire is a 16-item questionnaire on concussion symptom severity. Participants rate their symptoms (e.g. headache, dizziness, nausea) on a scale of 0 (not experienced at all) to 4 (a severe problem). Total scores range from 0 to 64, with higher scores indicating a worse outcome.
  units on a scale |  | 19.43 (14.11) | 20.67 (13.63) | 2.06 (4.19) | 14.1 (9.99)
GAD [Mean (Standard Deviation); unit: units on a scale] — The Generalized Anxiety Disorder is a 7-item questionnaire that assesses participant anxiety. Participants rate their experiences of the questions (e.g. feeling nervous, anxious, or on-edge) on a scale of 0 (not at all) to 3 (nearly every day). Total scores range from 0 to 21, with higher scores indicating worse outcomes.
  units on a scale |  | 10.89 (4.91) | 8.89 (5.37) | 3.43 (3.55) | 7.65 (4.57)
SDNN [Mean (Standard Deviation); unit: ms] — Standard deviation of the normal to normal interval (SDNN) is a measure that represents heart rate variability. An electrocardiogram was used to measure their SDNN for three minutes. Mean SDNN values were calculated. Higher SDNN values indicate improved autonomic function. Average SDNN for healthy individuals between 35 and 74 years of age are 37.9-45.7 ms (Dantas et al., 2017).
  ms |  | 43.86 (14.11) | 42.89 (16.6) | 46.29 (23.57) | 44.306 (17.99)
EEG [Mean (Standard Deviation); unit: Hz] — Electroencephalograph (EEG) values were calculated using z-scores of the EEG amplitude for frequencies between 2 and 30 Hz (0.1 Hz resolution) at all 47 Brodmann areas. Average mean deviations from normal values within the designated target Brodmann areas, at all frequencies (2-30 Hz), were calculated. Scores ranged from -3 to 3 standard deviations (measured in Hz). Increased deviation indicates a worse outcome.
  Hz |  | .4 (.95) | .07 (.43) | .5 (.82) | .31 (.67)

OUTCOME MEASURES:

1. Primary Outcome: Change In SDNN
Description: The interval between heartbeats, specifically the artifact-free intervals between R waves in the QRS complex, will be measured. This is known as the standard deviation of the norm (SDNN), and is a universal method of quantifying HRV (Camm et al., 1996). This information is collected using the Mindja application for android devices, created by Evoke Neuroscience.The physiologically relevant norms are a mean of 50 (SD 16) and a range from 32-93 ms (Shaffer F, Ginsberg JP. An Overview of Heart Rate variability Metrics and Norms. Frontiers in Public Health. 2017 Sep;5(258):1.)
Time Frame: baseline and post-intervention (8 weeks)
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Heart Rate Variability/Neurofeedback | Post-Concussed Control Group | Non-Concussed Control Group
Number analyzed (Participants) | 7 | 9 | 8
ms | 43. (12.1) | 21.87 (4.67) | 19.4 (4.4)

2. Primary Outcome: Number of Participants Making Driving Simulator Mistakes
Description: Participants will perform a driving simulation task using the DriveSafety CDS-250 driving simulator. It will record the performance, and afterwards a trained rater will review and evaluate the number of driving errors using a standardized assessment form. The number of individuals that made a driving simulator mistake are reported. The minimum is zero and the maximum is the number of participants in the Arm/Group. We are not aware of any physiologically relevant ranges for this measure.
Time Frame: baseline and post-intervention (8 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Heart Rate Variability/Neurofeedback | Post-Concussed Control Group | Non-Concussed Control Group
Number analyzed (Participants) | 7 | 9 | 8
Participants | 0 | 2 | 0

3. Primary Outcome: Change In Electrocardiograph Amplitudes
Description: The amplitude and power of alpha, beta, theta, and delta frequencies will be evaluated relative to reference norms (Gevensleben et al., 2010) and expressed as Z-scores (deviation from the mean divided by the standard deviation). In terms of physiologically relevant norms, 99% of the population will have scores between -3 and +3. This information is collected and stored in a secured cloud between Evoke Neuroscience and Western University.
Time Frame: baseline and post-intervention (8 weeks)
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Heart Rate Variability/Neurofeedback | Post-Concussed Control Group | Non-Concussed Control Group
Number analyzed (Participants) | 7 | 9 | 8
Z-score | -.23 (.64) | .33 (.79) | .87 (1.01)

4. Secondary Outcome: Change In Number and Severity of Post-concussive Symptoms
Description: These are assessed using the Rivermead Post Concussion Questionnaire (RPQ). It evaluates the severity of 16 common post-concussion symptoms over the past 24 hours (with the option to add 2 additional symptoms not already listed). Some examples include headache, sleep disturbance, noise sensitivity and blurred vision. It asks the evaluator to compare each symptom to how they would "normally" have felt prior to the concussion. It is a 5-point scale, which goes from 0-4. When the symptom is not experienced at all, the evaluator is to put a 0 (better outcome), whereas 4 indicates the symptom is a severe problem (worse outcome). Scores range from 0-72, where 72 represents experiencing all symptoms, and they are all a severe problem (worse outcome).
Time Frame: baseline and post-intervention (8 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Heart Rate Variability/Neurofeedback | Post-Concussed Control Group | Non-Concussed Control Group
Number analyzed (Participants) | 7 | 9 | 8
units on a scale | 18.36 (14.24) | 20.56 (14.56) | 1.5 (3.69)

5. Secondary Outcome: Change In Anxiety
Description: This is assessed using the Generalized Anxiety Disorder 7-Item Scale (GAD-7). Seven anxiety symptoms experienced over the past 2 weeks are evaluated on a 4-point scale, which goes from 0-3. Some examples include feeling nervous or anxious, inability to stop worrying, and trouble relaxing. When the symptom is not experienced at all, the evaluator is to put a 0 (better outcome), whereas 3 indicates the symptom is experienced nearly every day (worse outcome). Score totals range from 0 to 21, where 21 represents experiencing all symptoms, and they are all experienced nearly every day (worse outcome).
Time Frame: baseline and post-intervention (8 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Heart Rate Variability/Neurofeedback | Post-Concussed Control Group | Non-Concussed Control Group
Number analyzed (Participants) | 7 | 9 | 8
units on a scale | 8.56 (5.13) | 8.33 (6.04) | 2 (1.63)

ADVERSE EVENTS:
Time Frame: during the 8 week intervention
Arm/Group | Heart Rate Variability/Neurofeedback | Post-Concussed Control Group | Non-Concussed Control Group
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 0/7 | 0/9 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT03338036/Prot_SAP_000.pdf